CLINICAL TRIAL: NCT03788967
Title: A Phase 3, Randomized, Double-blind, Double-dummy, Multicenter, Prospective Study to Assess the Efficacy, Safety and Pharmacokinetics of Orally Administered Tebipenem Pivoxil Hydrobromide (SPR994) Compared to Intravenous Ertapenem in Patients With Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)
Brief Title: Study to Assess the Efficacy, Safety and Pharmacokinetics of Orally Administered Tebipenem Pivoxil Hydrobromide (SPR994) Compared to Intravenous Ertapenem in Participants With Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)
Acronym: ADAPT-PO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR994-301; 2018-003671-35 (EudraCT Number)
Record Dates: First submitted 2018-12-22; First posted 2018-12-28 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-06

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis
Keywords: Complicated Urinary Tract Infection; Acute Pyelonephritis
MeSH Terms: interventions — tebipenem; Ertapenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TBPM-PI-HBr 600 mg (Experimental): TBPM-PI-HBr 600 mg (300 mg×2 ) film-coated tablets, administered orally three times per day (every 8 hours [q8h] ± 0.5 h) plus a single dummy IV infusion over 30 minutes (min) once daily (every 24 hours [q24h] ± 0.5 h) up to Day 15; participants with moderate renal insufficiency (creatinine clearance [CrCl] >30 to ≤50 mL/min) required TBPM-PI-HBr dosage adjustment to 300 mg (one tablet) q8h ± 0.5 h.
  Interventions: Drug: TBPM-PI-HBr; Drug: Dummy Infusion
- Ertapenem 1 g (Active Comparator): Ertapenem for IV injection, administered as a 1-gram IV infusion over 30 min once daily (q24h ± 0.5 h) plus dummy placebo tablets administered orally q8h (±0.5 h) up to Day 14; no dose adjustment of ertapenem was required for participants with renal insufficiency.
  Interventions: Drug: Ertapenem; Drug: Dummy tablets

INTERVENTIONS:
Drug: TBPM-PI-HBr — TBPM-PI-HBr tablets administered orally.
  Other Names: SPR994
  Arms: TBPM-PI-HBr 600 mg
Drug: Ertapenem — Antibiotic Therapy for cUTI.
  Arms: Ertapenem 1 g
Drug: Dummy Infusion — Dummy intravenous infusion.
  Arms: TBPM-PI-HBr 600 mg
Drug: Dummy tablets — Dummy tablets orally.
  Arms: Ertapenem 1 g

SUMMARY:
The key purpose of this study is to evaluate the efficacy, safety and pharmacokinetics (PK) of tebipenem pivoxil hydrobromide (TBPM-PI-HBr) compared to intravenous (IV) ertapenem, in participants with complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP).

ELIGIBILITY:
Inclusion Criteria

1. Male and female participants at least 18 years of age.
2. Able to provide informed consent.
3. Able to ingest oral tablets for the anticipated treatment duration. If present at baseline, nausea and/or vomiting should have been mild or well-controlled with antiemetic therapy, in order to tolerate oral study drug.
4. Have a diagnosis of cUTI or AP as defined below:

   a. cUTI definition:

   At least Two of the following signs and symptoms:

   i. Chills, rigors, or fever; fever must be observed and documented by a health care provider (oral, tympanic, rectal or core temperature >38.0°C [>100.4°F])

   ii. Dysuria, urgency to void, or increased urinary frequency

   iii. Nausea or vomiting, as reported by the participants

   iv. Lower abdominal, suprapubic, or pelvic pain

   And at least One of the following risk factors for cUTI:

   i. Implanted urinary tract instrumentation (e.g., nephrostomy tube, ureteric stents, or other urinary tract prosthetic material), ongoing intermittent bladder catheterization, or presence of an indwelling bladder catheter (Note: bladder catheters that have been in place for >24 hours prior to Screening must be removed or replaced prior to collection of the Screening urine for urinalysis and culture, unless removal or replacement is considered unsafe or contraindicated).

   ii. Current known functional or anatomical abnormality of the urogenital tract, including anatomic abnormalities of the urinary tract, neurogenic bladder, or post-void residual urine volume of ≥ 100 mL within the past 6 months.

   iii. Complete or partial obstructive uropathy (e.g., nephrolithiasis, tumor, fibrosis, urethral stricture) that is expected to be medically or surgically treated during study drug therapy (prior to end of the treatment [EOT]).

   iv. Known intrinsic renal disease with blood urea nitrogen (BUN) >20 mg/deciliter (dL), or blood urea >42.8 mg/dL, or serum creatinine (Cr) >1.4 mg/dL.

   v. Urinary retention, including urinary retention in men due to previously diagnosed benign prostatic hyperplasia (BPH).

   b. AP definition: Acute flank pain (onset within 7 days prior to randomization) or costovertebral angle tenderness on physical examination.

   And at least One of the following signs and symptoms:

   i. Chills, rigors, or fever; fever must be observed and documented by a health care provider (oral, tympanic, rectal or core temperature >38.0°C [>100.4°F]).

   ii. Peripheral white blood cell count (WBC) >10,000/mm3 or bandemia (≥15% immature polymorphonuclear neutrophils (PMNs), regardless of WBC count).

   iii. Nausea or vomiting, as reported by the participants.

   iv. Dysuria, urgency to void, or increased urinary frequency.

   Note: Participants who meet the definition for cUTI (Inclusion Criterion 4a) and also have flank pain or costovertebral tenderness should be randomized as cUTI rather than AP.
5. Have an adequate urine specimen for evaluation and culture obtained within 24 h prior to randomization with evidence of pyuria that includes at least one of the following:

   1. At least 10 WBCs per high power field (hpf) in urine sediment.
   2. At least 10 WBCs per cubic millimeter (mm3) in unspun (non-centrifuged) urine.
   3. Positive leukocyte esterase (LE) on urinalysis. Note: Participants could be randomized and administered investigational product (IP) prior to knowledge of urine culture results.
6. Expectation, in the judgment of the Investigator, that the participant would survive with effective antibiotic therapy and appropriate supportive care for the anticipated duration of the study.
7. Willing to comply with all the study activities and procedures throughout the duration of the study.
8. Participants were required to use a highly-effective method of birth control; male participants were required to use an effective barrier method of contraception from Screening through LFU and for 90 days following the last dose if sexually active with a female of childbearing potential (FOCP); female participants must not have been pregnant or nursing, and were required to commit to either sexual abstinence or use at least two medically accepted, effective methods of birth control (e.g., condom, spermicidal gel, oral contraceptive, indwelling intrauterine device, hormonal implant/patch, injections, approved cervical ring) from Screening through LFU and for 90 days following the last dose.

Exclusion Criteria

1. Presence of any known or suspected disease or condition that, in the opinion of the Investigator, may have confounded the assessment of efficacy, including but not limited to the following:

   1. Perinephric or renal corticomedullary abscess.
   2. Uncomplicated urinary tract infection (cUTI) - (acute cystitis that does not meet the cUTI disease definition, see Inclusion Criterion 4a).
   3. Polycystic kidney disease.
   4. Recent history of trauma to the pelvis or urinary tract.
   5. Confirmed or suspected acute or chronic bacterial prostatitis, orchitis, or epididymitis.
   6. Chronic vesicoureteral reflux.
   7. Previous or planned renal transplantation.
   8. Previous or planned cystectomy or ileal loop surgery.
   9. Known or suspected non-renal source of infection (e.g., infective endocarditis, osteomyelitis, meningitis, pneumonia).
   10. Confirmed or suspected infection that is caused by a pathogen that is resistant to either IP (e.g., carbapenem-resistant pathogen), including infection caused by fungi (e.g., candiduria) or mycobacteria (e.g., urogenital tuberculosis).
2. Gross hematuria requiring intervention other than administration of IP or removal/placement of urinary tract instrumentation.
3. Urinary tract surgery within 7 days prior to randomization or urinary tract surgery planned during the study period (except surgery required relieving an obstruction or placing urinary tract instrumentation).
4. Creatinine clearance (CrCl) of ≤30 mL/min, as estimated by the Cockcroft-Gault formula:

   estimated Creatinine Clearance (eC_Cr) [mL/min]=((140-Age [yrs]) × Body Weight [kg] × [0.85 if Female])/(72 × Serum Creatinine [mg⁄dL]).
5. Anticipated concomitant use of non-study antibacterial drug therapy between randomization and the LFU Visit that would potentially effect outcome evaluations of cUTI/ AP, including but not limited to antibacterials with potential activity versus uropathogens, antibacterial drug prophylaxis, and antibacterial bladder irrigation.
6. Anticipated concomitant use of gastric acid-reducing medications between randomization and end-of-treatment (EOT), including proton pump inhibitors, histamine-2 receptor antagonists, and antacids.
7. Receipt of more than a single dose of a short-acting potentially effective antibiotic started within 72 h prior to randomization.

   Exception: Participants who received more than a single dose of short-acting potentially effective antibiotic within 72 h prior to randomization may be eligible for enrollment if they meet all of the following criteria:
   1. In the opinion of the Investigator they have failed the prior antibiotic therapy (e.g., have worsening signs and symptoms of cUTI/AP).
   2. Had a documented uropathogen (growth in urine culture >10^5 CFU/mL) that is resistant to the prior antibiotic therapy.
   3. Had a documented uropathogen that is carbapenem-susceptible.
   4. Received approval from the Medical Monitor to enroll the participants.
8. Severe hepatic impairment at Screening, as evidenced by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5x upper limit of normal (ULN) or total bilirubin >3x ULN, or clinical signs of cirrhosis or end-stage hepatic disease (e.g., ascites, hepatic encephalopathy).
9. Any signs of severe sepsis, including shock or profound hypotension defined as systolic blood pressure <90 mmHg or a decrease of >40 mmHg from baseline that is not responsive to fluid challenge.
10. Pregnant or breastfeeding women.
11. History of epilepsy or known seizure disorder (excluding a history of childhood febrile seizures).
12. Receipt of any investigational medication during the last 30 days or 5 half-lives, whichever is longer, prior to randomization.
13. Known history of human immunodeficiency virus (HIV) infection and or acquired immunodeficiency syndrome (AIDS)-defining illness, or known history of HIV infection and known CD4 count <200/mm^3 within the past year.
14. Presence of immunodeficiency or an immunocompromised condition including neutropenia (<1,000 neutrophils/mm^3 obtained from the local laboratory at Screening), hematologic malignancy, bone marrow transplant, or receiving immunosuppressive therapy such as cancer chemotherapy, medications for the rejection of transplantation, and long-term use of systemic corticosteroids (e.g., ≥20 mg/day of prednisone or systemic equivalent for at least 2 weeks).
15. A mean QT interval corrected using Fridericia's formula (QTcF) >480 msec based on triplicate ECGs at Screening.
16. History of significant hypersensitivity or allergic reaction to β-lactam antibiotics (e.g., cephalosporins, penicillins, carbapenems), product excipients (mannitol, microcrystalline cellulose, crospovidone, magnesium stearate, colloidal silicon dioxide, and Opadry®) or any contraindication to the use of ertapenem.
17. History of known genetic metabolism anomaly associated with carnitine deficiency (e.g., carnitine transporter defect, methylmalonic aciduria, propionic acidemia)
18. Requirement for concomitant use of valproic acid, divalproex sodium, or probenecid between randomization and EOT.
19. Unable or unwilling to comply with the protocol.
20. An employee of the Investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as a family member of the employee or the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1372 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MD, Study Director — Spero Therapeutics Inc
Locations (71):
- United States (2):
  - Medical Facility, La Mesa, California
  - Medical Facility, Miami, Florida
- Bulgaria (6):
  - Medical Facility, Blagoevgrad
  - Medical Facility, Dobrich
  - Medical Facility, Rousse
  - Medical Facility, Shumen
  - Medical Facility, Sofia
  - Medical Facility, Veliko Tarnovo
- Czechia (5):
  - Medical Facility, Karlovy Vary
  - Medical Facility, Liberec
  - Medical Facility, Prague
  - Medical Facility, Ústí nad Labem
  - Medical Facility, Zlín
- Estonia (3):
  - Medical Facility, Kohtla-Järve
  - Medical Facility, Tallinn
  - Medical Facility, Võru
- Georgia (2):
  - Medical Facility, Tbilisi
  - Medical Facility, Zestaponi
- Hungary (4):
  - Medical Facility, Budapest
  - Medical Facility, Nagykanizsa
  - Medical Facility, Nyíregyháza
  - Medical Facility, Tatabánya
- Latvia (2):
  - Medical Facility, Riga
  - Medical Facility, Valmiera
- Medical Facility, Chisinau, Moldova
- Poland (5):
  - Medical Facility, Katowice
  - Medical Facility, Krakow
  - Medical Facility, Lodz
  - Medical Facility, Oświęcim
  - Medical Facility, Wroclaw
- Romania (4):
  - Medical Facility, Bucharest
  - Medical Facility, Craiova
  - Medical Facility, Iași
  - Medical Facility, Oradea
- Russia (9):
  - Medical Facility, Arkhangelsk
  - Medical Facility, Lomonosov
  - Medical Facility, Penza
  - Medical Facility, Pyatigorsk
  - Medical Facility, Saint Petersburg
  - Medical facility, Saint Petersburg
  - Medical Facility, Smolensk
  - Medical Facility, Vsevolozhsk
  - Medical Facility, Yaroslavl
- Serbia (4):
  - Medical Facility, Belgrade
  - Medical Facility, Kragujevac
  - Medical Facility, Novi Sad
  - Medical Facility, Vršac
- Slovakia (6):
  - Medical Facility, Bratislava
  - Medical Facility, Galanta
  - Medical Facility, Lučenec
  - Medical Facility, Martin
  - Medical Facility, Poprad
  - Medical Facility, Svidník
- South Africa (6):
  - Medical Facility, Benoni
  - Medical Facility, Chatsworth
  - Medical Facility, Durban
  - Medical Facility, Johannesburg
  - Medical Facility, Middelburg
  - Medical Facility, Pretoria
- Ukraine (12):
  - Medical Facility, Cherkasy
  - Medical Facility, Chernihiv
  - Medical Facility, Dnipro
  - Medical Facility, Ivano-Frankivsk
  - Medical Facility, Kharkiv
  - Medical Facility, Lviv
  - Medical Facility, Mykolaiv
  - Medical Facility, Odesa
  - Medical Facility, Uzhhorod
  - Medical Facility, Vinnytsia
  - Medical Facility, Zaporizhia
  - Medical Facility, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eckburg PB, Muir L, Critchley IA, Walpole S, Kwak H, Phelan AM, Moore G, Jain A, Keutzer T, Dane A, Melnick D, Talley AK. Oral Tebipenem Pivoxil Hydrobromide in Complicated Urinary Tract Infection. N Engl J Med. 2022 Apr 7;386(14):1327-1338. doi: 10.1056/NEJMoa2105462. PMID 35388666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 95 study centers in Bulgaria, Czech Republic, Estonia, Georgia, Hungary, Latvia, Moldova, Poland, Romania, Russia, Serbia, Slovakia, South Africa, Ukraine, and the United States from 03 June 2019 to 27 May 2020.
Pre-assignment Details: Participants with diagnosis of complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP) were enrolled to receive tebipenem pivoxil hydrobromide (TBPM-PI-HBr) and ertapenem.
Period: Overall Study
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Started | 685 | 687
Micro-Intent-to-Treat (ITT) Population (Micro-ITT=all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens.) | 449 | 419
Completed | 653 | 663
Not Completed | 32 | 24
Not completed — Lost to Follow-up | 14 | 10
Not completed — Participant Non-Compliance/Uncooperativeness | 3 | 6
Not completed — Participant Withdrawal of Consent | 13 | 5
Not completed — Adverse Event | 1 | 1
Not completed — COVID-19 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g | Total
Number analyzed (Participants) | 685 | 687 | 1372
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (18.68) | 57.2 (18.23) | 56.9 (18.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 368 | 389 | 757
  Male | 317 | 298 | 615
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 5 | 18
  Not Hispanic or Latino | 672 | 682 | 1354
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 676 | 677 | 1353
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (Combined Clinical Cure and Microbiological Eradication) at Test-of-Cure (TOC) in Micro Intent-to-Treat Population
Description: Overall response is participants with combined clinical cure and microbiological eradication. Clinical cure is defined as complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted. Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 colony forming unit/milliliter (CFU/mL) and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline.
Time Frame: Day 19 (TOC)
Population: Microbiological intent-to-treat population (Micro-ITT) included all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
Participants | 264 | 258
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Non-Inferiority — The non-inferiority hypothesis test was a 1-sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the 95% CI for the difference in overall response was greater than -12.5%, non-inferiority was declared; Risk Difference = -3.3, 95% CI 2-sided [-9.7 to 3.2]

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) in The Safety Population
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a subject or clinical investigation participant administered a pharmaceutical product, which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational/experimental) product, whether or not related to this product.
Time Frame: From the first dose of administration up to Day 25 post-treatment ± 2 days (up to approximately 27 days)
Population: Safety analysis population included all randomized participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 685 | 687
Participants | 176 | 176

3. Secondary Outcome: Overall Response (Combined Clinical Cure Plus Microbiological Eradication) At Test-Of-Cure (TOC) In The Microbiologically Evaluable (ME) - TOC Population
Description: Overall response is participants with combined clinical cure and microbiological eradication. Clinical cure is defined as complete resolution or significant improvement of signs and symptoms of cUTI or acute pyelonephritis (AP) that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted. Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline.
Time Frame: Day 19 (TOC)
Population: Microbiologically evaluable (ME) - TOC is a subset which included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the evaluability review plan (ERP).
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 413 | 376
Participants | 254 | 247
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = -4.7, 95% CI 2-sided [-11.3 to 1.9]

4. Secondary Outcome: Clinical Cure at End-of-Treatment (EOT), TOC, and Sustained Clinical Cure at Late Follow-Up (LFU) Days in the Micro-ITT Populations
Description: Clinical cure is defined as number of participants with complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted. Sustained clinical cure is defined as participants who met criteria for clinical cure at TOC and remained free of signs and symptoms of cUTI or AP at LFU.
Time Frame: Days 15 (EOT), Day 19 (TOC) and Day 25 (LFU)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
Participants
  EOT | 446 | 410
  TOC | 418 | 392
  LFU | 398 | 377
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Statistical Analysis 1 (EOT); Test type: Other; Risk Difference = 1.4, 95% CI 2-sided [-0.1 to 3.4]
Statistical Analysis 2: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Statistical Analysis 2 (TOC); Test type: Other; Risk Difference = -0.6, 95% CI 2-sided [-4 to 2.8]
Statistical Analysis 3: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Statistical Analysis 3 (LFU); Test type: Other; Risk Difference = -1.5, 95% CI 2-sided [-5.7 to 2.6]

5. Secondary Outcome: Clinical Cure at EOT Days the Clinically Evaluable (CE-EOT) Populations
Description: Clinical cure is defined as number of participants with complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted.
Time Frame: Day 15 (EOT)
Population: CE-EOT population is a subset which included participants who meet the definition for the ITT population, have no important protocol deviations that would affect the assessment of efficacy, and had an outcome assessed as clinical cure or clinical failure at EOT.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 677 | 674
Participants | 673 | 665
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = 0.7, 95% CI 2-sided [-0.3 to 2.0]

6. Secondary Outcome: Clinical Cure at TOC in the CE-TOC Populations
Description: as for outcome 5
Time Frame: Day 19 (TOC)
Population: CE-TOC population is a subset which included participants who meet the definition for the ITT population, have no important protocol deviations that would affect the assessment of efficacy, and had an outcome assessed as clinical cure or clinical failure at TOC.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 641 | 637
Participants | 611 | 617
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = -1.6, 95% CI 2-sided [-3.8 to 0.6]

7. Secondary Outcome: Sustained Clinical Cure at LFU in the CE-LFU Populations
Description: Clinical cure is defined as number of participants with complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted. Sustained clinical cure is defined as number of participants who met criteria for clinical cure at TOC and remained free of signs and symptoms of cUTI or AP at LFU.
Time Frame: Day 25 (LFU)
Population: CE-LFU population is a subset which included participants who meet the definition for the ITT population, have no important protocol deviations that would affect the assessment of efficacy, and had an outcome assessed as clinical cure or clinical failure at LFU.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 596 | 596
Participants | 556 | 559
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = -0.5, 95% CI 2-sided [-3.3 to 2.3]

8. Secondary Outcome: Clinical Cure at EOT in the ME-EOT Populations
Description: as for outcome 5
Time Frame: Day 15 (EOT)
Population: ME-EOT population is a subset which included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the ERP.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 439 | 401
Participants | 437 | 394
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = 1.3, 95% CI 2-sided [-0.2 to 3.2]

9. Secondary Outcome: Clinical Cure at TOC Days in the ME-TOC Populations
Description: as for outcome 5
Time Frame: Day 19 (TOC)
Population: ME-TOC population is a subset which included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the ERP.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 413 | 376
Participants | 390 | 363
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = -2.2, 95% CI 2-sided [-5.3 to 0.8]

10. Secondary Outcome: Sustained Clinical Cure at LFU in the ME-LFU Population
Description: as for outcome 4
Time Frame: Day 25 (LFU)
Population: ME-LFU population is a subset which included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the ERP.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 391 | 353
Participants | 360 | 329
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = -1.2, 95% CI 2-sided [-5.1 to 2.6]

11. Secondary Outcome: By-Patient Microbiological Eradication at EOT, TOC, and Sustained Microbiological Eradication at LFU Days in the Micro-ITT Population
Description: Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline. Microbiological eradication is defined as number of participants with reduction of Baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at Baseline. Sustained Microbiological Eradication is defined as number of participants with microbiologic eradication at the TOC and no subsequent urine culture after TOC demonstrating recurrence of the original baseline uropathogen at ≥10^5 CFU/mL.
Time Frame: Days 15 (EOT), 19 (TOC) and 25 (LFU)
Population: Micro-ITT include all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
Participants
  EOT | 439 | 403
  TOC | 267 | 266
  LFU | 257 | 244
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Statistical Analysis 1 (EOT); Test type: Other; Risk Difference = 1.5, 95% CI 2-sided [-0.8 to 4.1]
Statistical Analysis 2: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Statistical Analysis 2 (TOC); Test type: Other; Risk Difference = -4.5, 95% CI 2-sided [-10.8 to 1.9]
Statistical Analysis 3: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = -1.5, 95% CI 2-sided [-7.9 to 5]

12. Secondary Outcome: By-Pathogen Microbiological Eradication Rate at EOT in the Micro-ITT Population
Description: Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline. Microbiological eradication rate is the percentage of pathogens being eradicated from the overall number of pathogens analyzed.
Time Frame: Days 15 (EOT)
Population: Micro-ITT-all randomized participants with confirmed diagnosis of cUTI/AP and positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens. Overall Number of Units Analyzed=number of pathogens available for analysis at given timepoint. Participant may have had more than 1 pathogen. Multiple isolates of same species/category from same participant are counted only once towards total.
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: Pathogens
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
Number analyzed (Pathogens) | 493 | 455
percentage of pathogen eradication
  Enterobacterales, Citrobacter braakii: number analyzed (Pathogens) | 0 | 2
  Enterobacterales, Citrobacter braakii |  | 100
  Enterobacterales, Citrobacter freundii: number analyzed (Pathogens) | 4 | 3
  Enterobacterales, Citrobacter freundii | 75.0 | 66.7
  Enterobacterales, Citrobacter koseri: number analyzed (Pathogens) | 3 | 4
  Enterobacterales, Citrobacter koseri | 100 | 100
  Enterobacterales, Enterobacter amnigenus: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter amnigenus |  | 100
  Enterobacterales, Enterobacter asburiae: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter asburiae |  | 100
  Enterobacterales, Enterobacter bugandensis: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter bugandensis |  | 100
  Enterobacterales, Enterobacter cloacae: number analyzed (Pathogens) | 11 | 8
  Enterobacterales, Enterobacter cloacae | 90.9 | 100
  Enterobacterales, Escherichia coli: number analyzed (Pathogens) | 287 | 270
  Enterobacterales, Escherichia coli | 98.3 | 96.7
  Enterobacterales, Klebsiella aerogenes: number analyzed (Pathogens) | 1 | 1
  Enterobacterales, Klebsiella aerogenes | 100 | 0.0
  Enterobacterales, Klebsiella oxytoca: number analyzed (Pathogens) | 4 | 3
  Enterobacterales, Klebsiella oxytoca | 100 | 100
  Enterobacterales, Klebsiella pneumoniae: number analyzed (Pathogens) | 53 | 71
  Enterobacterales, Klebsiella pneumoniae | 98.1 | 98.6
  Enterobacterales, Klebsiella variicola: number analyzed (Pathogens) | 2 | 4
  Enterobacterales, Klebsiella variicola | 100 | 100
  Enterobacterales, Morganella morganii: number analyzed (Pathogens) | 2 | 4
  Enterobacterales, Morganella morganii | 100 | 100
  Enterobacterales, Proteus hauseri: number analyzed (Pathogens) | 2 | 0
  Enterobacterales, Proteus hauseri | 100 |
  Enterobacterales, Proteus mirabilis: number analyzed (Pathogens) | 35 | 23
  Enterobacterales, Proteus mirabilis | 97.1 | 100
  Enterobacterales, Proteus penneri: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Proteus penneri |  | 100
  Enterobacterales, Proteus vulgaris: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Proteus vulgaris |  | 100
  Enterobacterales, Providencia rettgeri: number analyzed (Pathogens) | 4 | 3
  Enterobacterales, Providencia rettgeri | 100 | 100
  Enterobacterales, Providencia stuartii: number analyzed (Pathogens) | 1 | 1
  Enterobacterales, Providencia stuartii | 100 | 100
  Enterobacterales, Raoultella ornithinolytica: number analyzed (Pathogens) | 2 | 0
  Enterobacterales, Raoultella ornithinolytica | 100 |
  Enterobacterales, Serratia liquefaciens: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Serratia liquefaciens |  | 100
  Enterobacterales, Serratia marcescens: number analyzed (Pathogens) | 4 | 2
  Enterobacterales, Serratia marcescens | 100 | 100
  Gram Positive, Enterococcus faecalis: number analyzed (Pathogens) | 58 | 36
  Gram Positive, Enterococcus faecalis | 94.8 | 91.7
  Gram Positive, Enterococcus faecium: number analyzed (Pathogens) | 5 | 2
  Gram Positive, Enterococcus faecium | 100 | 100
  Gram Positive, Enterococcus hirae: number analyzed (Pathogens) | 1 | 0
  Gram Positive, Enterococcus hirae | 100 |
  Gram Positive, Staphylococcus aureus: number analyzed (Pathogens) | 5 | 8
  Gram Positive, Staphylococcus aureus | 100 | 75.0
  Gram Positive, Staphylococcus lugdunensis: number analyzed (Pathogens) | 2 | 1
  Gram Positive, Staphylococcus lugdunensis | 100 | 100
  Gram Positive, Staphylococcus saprophyticus: number analyzed (Pathogens) | 4 | 6
  Gram Positive, Staphylococcus saprophyticus | 100 | 100
  Gram Positive, Streptococcus gallolyticus: number analyzed (Pathogens) | 1 | 0
  Gram Positive, Streptococcus gallolyticus | 100 |

13. Secondary Outcome: By-Pathogen Microbiological Eradication Rate at TOC in the Micro-ITT Population
Description: as for outcome 12
Time Frame: Day 19 (TOC)
Population: Micro-ITT included all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens. Number analyzed are the number of pathogens available for analysis at the given timepoint.
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: Pathogens
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
Number analyzed (Pathogens) | 493 | 455
percentage of pathogen eradication
  Enterobacterales, Citrobacter braakii: number analyzed (Pathogens) | 0 | 2
  Enterobacterales, Citrobacter braakii |  | 100
  Enterobacterales, Citrobacter freundii: number analyzed (Pathogens) | 4 | 3
  Enterobacterales, Citrobacter freundii | 50.0 | 100
  Enterobacterales, Citrobacter koseri: number analyzed (Pathogens) | 3 | 4
  Enterobacterales, Citrobacter koseri | 66.7 | 50.0
  Enterobacterales, Enterobacter amnigenus: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter amnigenus |  | 100
  Enterobacterales, Enterobacter asburiae: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter asburiae |  | 100
  Enterobacterales, Enterobacter bugandensis: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter bugandensis |  | 100
  Enterobacterales, Enterobacter cloacae: number analyzed (Pathogens) | 11 | 8
  Enterobacterales, Enterobacter cloacae | 54.5 | 50.0
  Enterobacterales, Escherichia coli: number analyzed (Pathogens) | 287 | 270
  Enterobacterales, Escherichia coli | 62.7 | 65.2
  Enterobacterales, Klebsiella aerogenes: number analyzed (Pathogens) | 1 | 1
  Enterobacterales, Klebsiella aerogenes | 0.0 | 0.0
  Enterobacterales, Klebsiella oxytoca: number analyzed (Pathogens) | 4 | 3
  Enterobacterales, Klebsiella oxytoca | 75.0 | 33.3
  Enterobacterales, Klebsiella pneumoniae: number analyzed (Pathogens) | 53 | 71
  Enterobacterales, Klebsiella pneumoniae | 45.3 | 63.4
  Enterobacterales, Klebsiella variicola: number analyzed (Pathogens) | 2 | 4
  Enterobacterales, Klebsiella variicola | 50.0 | 75.0
  Enterobacterales, Morganella morganii: number analyzed (Pathogens) | 4 | 1
  Enterobacterales, Morganella morganii | 100 | 100
  Enterobacterales, Proteus hauseri: number analyzed (Pathogens) | 2 | 0
  Enterobacterales, Proteus hauseri | 100 |
  Enterobacterales, Proteus mirabilis: number analyzed (Pathogens) | 35 | 23
  Enterobacterales, Proteus mirabilis | 48.6 | 69.6
  Enterobacterales, Proteus penneri: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Proteus penneri |  | 100
  Enterobacterales, Proteus vulgaris: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Proteus vulgaris |  | 100
  Enterobacterales, Providencia rettgeri: number analyzed (Pathogens) | 4 | 3
  Enterobacterales, Providencia rettgeri | 100 | 100
  Enterobacterales, Providencia stuartii: number analyzed (Pathogens) | 1 | 1
  Enterobacterales, Providencia stuartii | 0.0 | 100
  Enterobacterales, Raoultella ornithinolytica: number analyzed (Pathogens) | 2 | 0
  Enterobacterales, Raoultella ornithinolytica | 100 |
  Enterobacterales, Serratia liquefaciens: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Serratia liquefaciens |  | 100
  Enterobacterales, Serratia marcescens: number analyzed (Pathogens) | 4 | 2
  Enterobacterales, Serratia marcescens | 50.0 | 100
  Gram Positive, Enterococcus faecalis: number analyzed (Pathogens) | 58 | 36
  Gram Positive, Enterococcus faecalis | 67.2 | 55.6
  Gram Positive, Enterococcus faecium: number analyzed (Pathogens) | 5 | 2
  Gram Positive, Enterococcus faecium | 100 | 100
  Gram Positive, Enterococcus hirae: number analyzed (Pathogens) | 1 | 0
  Gram Positive, Enterococcus hirae | 100 |
  Gram Positive, Staphylococcus aureus: number analyzed (Pathogens) | 5 | 8
  Gram Positive, Staphylococcus aureus | 100 | 37.5
  Gram Positive, Staphylococcus lugdunensis: number analyzed (Pathogens) | 2 | 1
  Gram Positive, Staphylococcus lugdunensis | 100 | 100
  Gram Positive, Staphylococcus saprophyticus: number analyzed (Pathogens) | 4 | 6
  Gram Positive, Staphylococcus saprophyticus | 100 | 83.3
  Gram Positive, Streptococcus gallolyticus: number analyzed (Pathogens) | 1 | 0
  Gram Positive, Streptococcus gallolyticus | 100 |

14. Secondary Outcome: By-Pathogen Sustained Microbiological Eradication Rate at LFU in the Micro-ITT Population (m-ITT)
Description: Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline. Sustained Microbiological Eradication is defined as microbiologic eradication at the TOC and no subsequent urine culture after TOC demonstrating recurrence of the original baseline uropathogen at ≥10^5 CFU/mL. Microbiological eradication rate is the percentage of pathogens being eradicated from the overall number of pathogen analyzed.
Time Frame: Day 25 (LFU)
Population: mITT-all randomized participants with confirmed diagnosis of cUTI/AP & positive Screening urine culture defined as growth of one/two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens. Overall Number of Units Analyzed are number of enterobacterale pathogens. Participant may have more than 1 pathogen. Multiple isolates of same species/category from same participants are counted once towards total.
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: Pathogens
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
Number analyzed (Pathogens) | 417 | 402
percentage of pathogen eradication
  Citrobacter braakii: number analyzed (Pathogens) | 0 | 2
  Citrobacter braakii |  | 100
  Citrobacter freundii: number analyzed (Pathogens) | 4 | 3
  Citrobacter freundii | 50.0 | 100
  Citrobacter koseri: number analyzed (Pathogens) | 4 | 3
  Citrobacter koseri | 66.7 | 50.0
  Enterobacter amnigenus: number analyzed (Pathogens) | 0 | 1
  Enterobacter amnigenus |  | 100
  Enterobacter asburiae: number analyzed (Pathogens) | 0 | 1
  Enterobacter asburiae |  | 0
  Enterobacter bugandensis: number analyzed (Pathogens) | 0 | 1
  Enterobacter bugandensis |  | 100
  Enterobacter cloacae: number analyzed (Pathogens) | 11 | 8
  Enterobacter cloacae | 54.5 | 37.5
  Enterococcus faecalis: number analyzed (Pathogens) | 58 | 36
  Enterococcus faecalis | 63.8 | 50.0
  Enterococcus faecium: number analyzed (Pathogens) | 5 | 2
  Enterococcus faecium | 100 | 100
  Enterococcus hirae: number analyzed (Pathogens) | 1 | 0
  Enterococcus hirae | 100 |
  Escherichia coli: number analyzed (Pathogens) | 287 | 270
  Escherichia coli | 59.9 | 60.0
  Klebsiella aerogenes: number analyzed (Pathogens) | 1 | 1
  Klebsiella aerogenes | 0.0 | 0.0
  Klebsiella oxytoca: number analyzed (Pathogens) | 4 | 3
  Klebsiella oxytoca | 75.0 | 33.3
  Klebsiella pneumoniae: number analyzed (Pathogens) | 53 | 71
  Klebsiella pneumoniae | 43.4 | 60.6
  Klebsiella variicola: number analyzed (Pathogens) | 2 | 4
  Klebsiella variicola | 50.0 | 75.0
  Morganella morganii: number analyzed (Pathogens) | 4 | 1
  Morganella morganii | 100 | 100
  Proteus hauseri: number analyzed (Pathogens) | 2 | 0
  Proteus hauseri | 100 |
  Proteus mirabilis: number analyzed (Pathogens) | 35 | 23
  Proteus mirabilis | 48.6 | 60.9
  Proteus penneri: number analyzed (Pathogens) | 0 | 1
  Proteus penneri |  | 100
  Proteus vulgaris: number analyzed (Pathogens) | 0 | 1
  Proteus vulgaris |  | 100
  Providencia rettgeri: number analyzed (Pathogens) | 4 | 3
  Providencia rettgeri | 100 | 100
  Providencia stuartii: number analyzed (Pathogens) | 1 | 1
  Providencia stuartii | 0.0 | 100
  Raoultella ornithinolytica: number analyzed (Pathogens) | 2 | 0
  Raoultella ornithinolytica | 100 |
  Serratia liquefaciens: number analyzed (Pathogens) | 0 | 1
  Serratia liquefaciens |  | 100
  Serratia marcescens: number analyzed (Pathogens) | 4 | 2
  Serratia marcescens | 50.0 | 100
  Staphylococcus aureus: number analyzed (Pathogens) | 5 | 8
  Staphylococcus aureus | 100 | 37.5
  Staphylococcus lugdunensis: number analyzed (Pathogens) | 2 | 1
  Staphylococcus lugdunensis | 100 | 100
  Staphylococcus saprophyticus: number analyzed (Pathogens) | 4 | 6
  Staphylococcus saprophyticus | 100 | 83.3
  Staphylococcus gallolyticus: number analyzed (Pathogens) | 1 | 0
  Staphylococcus gallolyticus | 100 |

15. Secondary Outcome: By-Patient Microbiological Eradication at EOT in the ME-EOT Populations
Description: Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline.
Time Frame: Day 15 (EOT)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 439 | 401
Participants | 436 | 399
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = -0.2, 95% CI 2-sided [-1.6 to 1.2]

16. Secondary Outcome: By-Patient Microbiological Eradication at TOC in the ME-TOC Population
Description: Microbiological eradication is defined as number of participants with reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline. Microbiological eradication rate is the percentage of pathogens being eradicated from the overall number of pathogens analyzed.
Time Frame: Day 15 (TOC)
Population: ME-TOC population included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the ERP.
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 413 | 376
Participants | 257 | 254
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = -5.9, 95% CI 2-sided [-12.4 to 0.7]

17. Secondary Outcome: By-Patient Sustained Microbiological Eradication at LFU Days in the ME-LFU Populations
Description: Microbiological eradication is defined as number of participants with reduction of baseline urine pathogen(s) to <10^3 colony forming unit/milliliter (CFU/mL) and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline. Sustained Microbiological Eradication is defined participants with microbiologic eradication at the TOC and no subsequent urine culture after TOC demonstrating recurrence of the original baseline uropathogen at ≥10^5 CFU/mL.
Time Frame: Day 25 (LFU)
Population: ME-LFU population included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the ERP
Measure: Count of Participants; unit: Participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 391 | 353
Participants | 234 | 216
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference (RD) = -1.6, 95% CI 2-sided [-8.5 to 5.3]

18. Secondary Outcome: By-pathogen Microbiological Eradication Rate in Participants at EOT in the ME-EOT Populations
Description: as for outcome 16
Time Frame: Day 15 (EOT)
Population: ME-EOT population included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the ERP. Number analyzed are the number of pathogens available for analysis at the given timepoint.
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: Pathogens
Groups:
- TBPM-PI-HBr: TBPM-PI-HBr 600 mg (300 mg×2 ) film-coated tablets, administered orally three times per day (every 8 hours [q8h] ± 0.5 h) plus a single dummy IV infusion over 30 minutes (min) once daily (every 24 hours [q24h] ± 0.5 h) up to Day 15; participants with moderate renal insufficiency (creatinine clearance [CrCl] >30 to ≤50 mL/min) required TBPM-PI-HBr dosage adjustment to 300 mg (one tablet) q8h ± 0.5 h.
- Ertapenem: Ertapenem for IV injection, administered as a 1-gram IV infusion over 30 min once daily (q24h ± 0.5 h) plus dummy placebo tablets administered orally q8h (±0.5 h) up to Day 14; no dose adjustment of ertapenem was required for participants with renal insufficiency.
Arm/Group | TBPM-PI-HBr | Ertapenem
Number analyzed (Participants) | 439 | 401
Number analyzed (Pathogens) | 481 | 436
percentage of pathogen eradication
  Enterobacterales, Citrobacter braakii: number analyzed (Pathogens) | 0 | 2
  Enterobacterales, Citrobacter braakii |  | 100
  Enterobacterales, Citrobacter freundii: number analyzed (Pathogens) | 3 | 2
  Enterobacterales, Citrobacter freundii | 100 | 100
  Enterobacterales, Citrobacter koseri: number analyzed (Pathogens) | 3 | 4
  Enterobacterales, Citrobacter koseri | 100 | 100
  Enterobacterales, Enterobacter amnigenus: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter amnigenus |  | 100
  Enterobacterales, Enterobacter asburiae: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter asburiae |  | 100
  Enterobacterales, Enterobacter bugandensis: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter bugandensis |  | 100
  Enterobacterales, Enterobacter cloacae: number analyzed (Pathogens) | 11 | 8
  Enterobacterales, Enterobacter cloacae | 90.9 | 100
  Enterobacterales, Escherichia coli: number analyzed (Pathogens) | 282 | 257
  Enterobacterales, Escherichia coli | 99.6 | 100
  Enterobacterales, Klebsiella aerogenes: number analyzed (Pathogens) | 1 | 0
  Enterobacterales, Klebsiella aerogenes | 100 |
  Enterobacterales, Klebsiella oxytoca: number analyzed (Pathogens) | 4 | 3
  Enterobacterales, Klebsiella oxytoca | 100 | 100
  Enterobacterales, Klebsiella pneumoniae: number analyzed (Pathogens) | 52 | 70
  Enterobacterales, Klebsiella pneumoniae | 100 | 100
  Enterobacterales, Klebsiella variicola: number analyzed (Pathogens) | 2 | 4
  Enterobacterales, Klebsiella variicola | 100 | 100
  Enterobacterales, Morganella morganii: number analyzed (Pathogens) | 4 | 1
  Enterobacterales, Morganella morganii | 100 | 100
  Enterobacterales, Proteus hauseri: number analyzed (Pathogens) | 2 | 0
  Enterobacterales, Proteus hauseri | 100 |
  Enterobacterales, Proteus mirabilis: number analyzed (Pathogens) | 34 | 23
  Enterobacterales, Proteus mirabilis | 100 | 100
  Enterobacterales, Proteus penneri: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Proteus penneri |  | 100
  Enterobacterales, Proteus vulgaris: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Proteus vulgaris |  | 100
  Enterobacterales, Providencia rettgeri: number analyzed (Pathogens) | 4 | 3
  Enterobacterales, Providencia rettgeri | 100 | 100
  Enterobacterales, Providencia stuartii: number analyzed (Pathogens) | 1 | 1
  Enterobacterales, Providencia stuartii | 100 | 100
  Enterobacterales, Raoultella ornithinolytica: number analyzed (Pathogens) | 2 | 0
  Enterobacterales, Raoultella ornithinolytica | 100 |
  Enterobacterales, Serratia liquefaciens: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Serratia liquefaciens |  | 100
  Enterobacterales, Serratia marcescens: number analyzed (Pathogens) | 4 | 2
  Enterobacterales, Serratia marcescens | 100 | 100
  Gram Positive, Enterococcus faecalis: number analyzed (Pathogens) | 54 | 34
  Gram Positive, Enterococcus faecalis | 98.1 | 97.1
  Gram Positive, Enterococcus faecium: number analyzed (Pathogens) | 5 | 2
  Gram Positive, Enterococcus faecium | 100 | 100
  Gram Positive, Enterococcus hirae: number analyzed (Pathogens) | 1 | 0
  Gram Positive, Enterococcus hirae | 100 |
  Gram Positive, Staphylococcus aureus: number analyzed (Pathogens) | 5 | 7
  Gram Positive, Staphylococcus aureus | 100 | 85.7
  Gram Positive, Staphylococcus lugdunensis: number analyzed (Pathogens) | 2 | 1
  Gram Positive, Staphylococcus lugdunensis | 100 | 100
  Gram Positive,Staphylococcus saprophyticus: number analyzed (Pathogens) | 4 | 6
  Gram Positive,Staphylococcus saprophyticus | 100 | 100
  Gram Positive, Streptococcus gallolyticus: number analyzed (Pathogens) | 1 | 0
  Gram Positive, Streptococcus gallolyticus | 100 |

19. Secondary Outcome: By-pathogen Microbiological Eradication Rate in Participants at TOC in the ME-TOC Populations
Description: Microbiological eradication is defined as number of participants with reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline. Microbiological eradication rate is the percentage of pathogens being eradicated from the overall number of participants analyzed.
Time Frame: Day 19 (TOC)
Population: ME-EOT population included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the ERP. Number analyzed are the number of pathogens available for analysis at the given timepoint. A participant may have had more than 1 pathogen. Multiple isolates of the same species/category from the same participants are counted only once towards total.
Measure: Number; unit: percentage of pathogen eradication
Units Other Than Participants: Pathogens
Arm/Group | TBPM-PI-HBr | Ertapenem
Number analyzed (Participants) | 413 | 376
Number analyzed (Pathogens) | 451 | 408
percentage of pathogen eradication
  Enterobacterales, Citrobacter braakii: number analyzed (Pathogens) | 0 | 2
  Enterobacterales, Citrobacter braakii |  | 100
  Enterobacterales, Citrobacter freundii: number analyzed (Pathogens) | 3 | 3
  Enterobacterales, Citrobacter freundii | 66.7 | 100
  Enterobacterales, Citrobacter koseri: number analyzed (Pathogens) | 3 | 3
  Enterobacterales, Citrobacter koseri | 66.7 | 66.7
  Enterobacterales, Enterobacter amnigenus: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter amnigenus |  | 100
  Enterobacterales, Enterobacter asburiae: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter asburiae |  | 100
  Enterobacterales, Enterobacter bugandensis: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Enterobacter bugandensis |  | 100
  Enterobacterales, Enterobacter cloacae: number analyzed (Pathogens) | 11 | 8
  Enterobacterales, Enterobacter cloacae | 54.5 | 50.0
  Enterobacterales, Escherichia coli: number analyzed (Pathogens) | 263 | 243
  Enterobacterales, Escherichia coli | 65.8 | 68.3
  Enterobacterales, Klebsiella aerogenes: number analyzed (Pathogens) | 1 | 0
  Enterobacterales, Klebsiella aerogenes | 0.0 |
  Enterobacterales, Klebsiella oxytoca: number analyzed (Pathogens) | 3 | 2
  Enterobacterales, Klebsiella oxytoca | 100 | 50.0
  Enterobacterales, Klebsiella pneumoniae: number analyzed (Pathogens) | 49 | 62
  Enterobacterales, Klebsiella pneumoniae | 49.0 | 71.0
  Enterobacterales, Klebsiella variicola: number analyzed (Pathogens) | 2 | 4
  Enterobacterales, Klebsiella variicola | 50.0 | 75.0
  Enterobacterales, Morganella morganii: number analyzed (Pathogens) | 4 | 1
  Enterobacterales, Morganella morganii | 100 | 100
  Enterobacterales, Proteus hauseri: number analyzed (Pathogens) | 2 | 0
  Enterobacterales, Proteus hauseri | 100 |
  Enterobacterales, Proteus mirabilis: number analyzed (Pathogens) | 31 | 21
  Enterobacterales, Proteus mirabilis | 51.6 | 76.2
  Enterobacterales, Proteus penneri: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Proteus penneri |  | 100
  Enterobacterales, Proteus vulgaris: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Proteus vulgaris |  | 100
  Enterobacterales, Providencia rettgeri: number analyzed (Pathogens) | 3 | 2
  Enterobacterales, Providencia rettgeri | 100 | 100
  Enterobacterales, Providencia stuartii: number analyzed (Pathogens) | 1 | 1
  Enterobacterales, Providencia stuartii | 0.0 | 100
  Enterobacterales, Raoultella ornithinolytica: number analyzed (Pathogens) | 2 | 0
  Enterobacterales, Raoultella ornithinolytica | 100 |
  Enterobacterales, Serratia liquefaciens: number analyzed (Pathogens) | 0 | 1
  Enterobacterales, Serratia liquefaciens |  | 100
  Enterobacterales, Serratia marcescens: number analyzed (Pathogens) | 3 | 2
  Enterobacterales, Serratia marcescens | 66.7 | 100
  Gram Positive, Enterococcus faecalis: number analyzed (Pathogens) | 53 | 33
  Gram Positive, Enterococcus faecalis | 69.8 | 57.6
  Gram Positive, Enterococcus faecium: number analyzed (Pathogens) | 5 | 2
  Gram Positive, Enterococcus faecium | 100 | 100
  Gram Positive, Enterococcus hirae: number analyzed (Pathogens) | 1 | 0
  Gram Positive, Enterococcus hirae | 100 |
  Gram Positive, Staphylococcus aureus: number analyzed (Pathogens) | 4 | 6
  Gram Positive, Staphylococcus aureus | 100 | 50.0
  Gram Positive, Staphylococcus lugdunensis: number analyzed (Pathogens) | 2 | 1
  Gram Positive, Staphylococcus lugdunensis | 100 | 100
  Gram Positive,Staphylococcus saprophyticus: number analyzed (Pathogens) | 4 | 6
  Gram Positive,Staphylococcus saprophyticus | 100 | 83.3
  Gram Positive, Streptococcus gallolyticus: number analyzed (Pathogens) | 1 | 0
  Gram Positive, Streptococcus gallolyticus | 100 |

20. Secondary Outcome: By-pathogen Sustained Microbiological Eradication Rate in Participants at LFU in the ME-LFU Populations
Description: Microbiological eradication is defined as number of participants with reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline. Sustained Microbiological Eradication is defined participants with microbiologic eradication at the TOC and no subsequent urine culture after TOC demonstrating recurrence of the original baseline uropathogen at ≥10^5 CFU/mL.Microbiological eradication rate is the percentage of pathogens being eradicated from the overall number of pathogen analyzed.
Time Frame: Day 25 (LFU)
Population: ME-LFU population included participants who met the definitions of both the micro-ITT Population and CE Population and were defined for each visit for the analyses in the ME Population at each respective visit as outlined in the ERP. Overall Number of Units Analyzed are the number of enterobacteral pathogens. A participant may have had more than 1 pathogen. Multiple isolates of the same species/category from the same participants are counted only once towards total.
Measure: Number; unit: percentage of pathogens eradications
Units Other Than Participants: Pathogens
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 391 | 353
Number analyzed (Pathogens) | 391 | 353
percentage of pathogens eradications
  Citrobacter braakii: number analyzed (Pathogens) | 0 | 2
  Citrobacter braakii |  | 100
  Citrobacter freundii: number analyzed (Pathogens) | 3 | 3
  Citrobacter freundii | 66.7 | 100
  Citrobacter koseri: number analyzed (Pathogens) | 2 | 3
  Citrobacter koseri | 100 | 66.7
  Enterobacter amnigenus: number analyzed (Pathogens) | 0 | 1
  Enterobacter amnigenus |  | 100
  Enterobacter asburiae: number analyzed (Pathogens) | 0 | 1
  Enterobacter asburiae |  | 0
  Enterobacter bugandensis: number analyzed (Pathogens) | 0 | 1
  Enterobacter bugandensis |  | 100
  Enterobacter cloacae: number analyzed (Pathogens) | 9 | 6
  Enterobacter cloacae | 55.6 | 33.3
  Enterococcus faecalis: number analyzed (Pathogens) | 51 | 34
  Enterococcus faecalis | 66.7 | 52.9
  Enterococcus faecium: number analyzed (Pathogens) | 5 | 2
  Enterococcus faecium | 100 | 100
  Enterococcus hirae: number analyzed (Pathogens) | 1 | 0
  Enterococcus hirae | 100 |
  Escherichia coli: number analyzed (Pathogens) | 250 | 228
  Escherichia coli | 62.4 | 61.8
  Klebsiella aerogenes: number analyzed (Pathogens) | 1 | 0
  Klebsiella aerogenes | 0 |
  Klebsiella oxytoca: number analyzed (Pathogens) | 2 | 2
  Klebsiella oxytoca | 100 | 50.0
  Klebsiella pneumoniae: number analyzed (Pathogens) | 45 | 57
  Klebsiella pneumoniae | 46.7 | 68.4
  Klebsiella variicola: number analyzed (Pathogens) | 2 | 3
  Klebsiella variicola | 50.0 | 66.7
  Morganella morganii: number analyzed (Pathogens) | 4 | 1
  Morganella morganii | 100 | 100
  Proteus hauseri: number analyzed (Pathogens) | 2 | 0
  Proteus hauseri | 100 |
  Proteus mirabilis: number analyzed (Pathogens) | 29 | 40
  Proteus mirabilis | 51.7 | 70.0
  Proteus penneri: number analyzed (Pathogens) | 0 | 1
  Proteus penneri |  | 100
  Proteus vulgaris: number analyzed (Pathogens) | 0 | 1
  Proteus vulgaris |  | 100
  Providencia rettgeri: number analyzed (Pathogens) | 3 | 3
  Providencia rettgeri | 100 | 100
  Providencia stuartii: number analyzed (Pathogens) | 1 | 1
  Providencia stuartii | 0.0 | 100
  Raoultella ornithinolytica: number analyzed (Pathogens) | 2 | 0
  Raoultella ornithinolytica | 100 |
  Serratia liquefaciens: number analyzed (Pathogens) | 0 | 1
  Serratia liquefaciens |  | 100
  Serratia marcescens: number analyzed (Pathogens) | 3 | 2
  Serratia marcescens | 66.7 | 100
  Staphylococcus aureus: number analyzed (Pathogens) | 4 | 6
  Staphylococcus aureus | 100 | 50.0
  1Staphylococcus lugdunensis: number analyzed (Pathogens) | 2 | 1
  1Staphylococcus lugdunensis | 100 | 100
  Staphylococcus saprophyticus: number analyzed (Pathogens) | 4 | 5
  Staphylococcus saprophyticus | 100 | 80.0
  Staphylococcus gallolyticus: number analyzed (Pathogens) | 1 | 0
  Staphylococcus gallolyticus | 100 |

21. Secondary Outcome: Overall Response Rate (Combined Clinical Cure Plus Microbiological Eradication) In Subgroup Including: Stratified Infection Category
Description: Overall response rate is percentage of participants with combined clinical cure plus microbiological eradication. Clinical cure is defined as complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted. Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 colony forming unit/milliliter (CFU/mL) and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline.
Time Frame: Day 19 (TOC)
Population: Micro-ITT population included all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens. Number analyzed are the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
percentage of participants
  AP: number analyzed (Participants) | 226 | 201
  AP | 65.9 | 70.6
  cUTI: number analyzed (Participants) | 223 | 218
  cUTI | 51.6 | 53.2
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Overall response for participants with AP; Test type: Other; Risk Difference = -4.7, 95% CI 2-sided [-13.5 to 4.1]
Statistical Analysis 2: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Overall response in participants with cUTI; Test type: Other; Risk Difference = -1.6, 95% CI 2-sided [-11.0 to 7.7]

22. Secondary Outcome: Overall Response Rate (Combined Clinical Cure Plus Microbiological Eradication) at TOC In Subgroup Stratified Age Category
Description: Overall response rate is percentage of participants with combined clinical cure plus microbiological eradication. Clinical cure is defined as complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted. Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 CFU/mL and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline.
Time Frame: Day 19 (TOC)
Population: Micro-ITT population included all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens. Number analyzed is number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
percentage of participants
  ≥18 to <65 years: number analyzed (Participants) | 246 | 222
  ≥18 to <65 years | 66.7 | 65.3
  ≥65 to <75 years: number analyzed (Participants) | 122 | 132
  ≥65 to <75 years | 49.2 | 57.6
  ≥75 years: number analyzed (Participants) | 81 | 65
  ≥75 years | 49.4 | 56.9
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; Risk Difference = 1.4, 95% CI 2-sided [-7.2 to 9.9]
Statistical Analysis 2: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; ≥65 to <75 years; Test type: Other; Risk Difference (RD) = -8.4, 95% CI 2-sided [-20.6 to 3.8]
Statistical Analysis 3: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; ≥75 years; Test type: Other; Risk Difference (RD) = -7.5, 95% CI 2-sided [-23.8 to 8.7]

23. Secondary Outcome: Overall Response Rate (Combined Clinical Cure Plus Microbiological Eradication) at TOC In Subgroup Including Region
Description: Overall response rate is percentage of participants with combined clinical cure plus microbiological eradication. Clinical cure is defined as complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted. Microbiological eradication is defined as reduction of baseline urine pathogen(s) to <10^3 colony forming unit/milliliter (CFU/mL) and negative repeated blood culture if blood culture was positive for uropathogen growth at baseline. The point estimate and confidence interval (CI) is presented for Central and eastern Europe subgroup.
Time Frame: Day 25 (LFU)
Population: Micro-ITT included all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens. Number analyzed is number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
percentage of participants
  Central and Eastern Europe: number analyzed (Participants) | 443 | 413
  Central and Eastern Europe | 58.9 | 62.0
  South Africa: number analyzed (Participants) | 3 | 2
  South Africa | 100 | 0.0
  United States: number analyzed (Participants) | 3 | 4
  United States | 0.0 | 50.0
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Central and Eastern Europe; Test type: Other; Risk Difference = -3.1, 95% CI 2-sided [-9.6 to 3.5]

24. Secondary Outcome: Time (Days) to Resolution or Improvement of Signs and Symptoms of cUTI and AP Present a Baseline in the Micro-ITT Populations
Description: Time (days) to resolution or improvement of signs and symptoms of cUTI and AP present at baseline was defined as follows: date of the first visit at which all baseline signs/symptoms have improved by at least 1 grade with worsening of none and development of no new signs/symptoms of the index infection minus the date of randomization.
Time Frame: Day 25 (LFU)
Population: Micro-ITT population included all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥105 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
days | 4.1 (3.85) | 3.7 (3.26)
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; p = 0.044, Log Rank

25. Secondary Outcome: Time (Days) to Defervescence in Micro-ITT Population With a Documented Fever at Screening or Day 1
Description: Time to Defervescence (days) = date of first post-baseline temperature measure with maximum daily Temperature ≤38°C at the date of randomization.
Time Frame: Day 25 (LFU)
Population: Micro-ITT population included all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens. Overall number of participants analyzed are the participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 226 | 193
days | 2.2 (1.33) | 2.2 (1.40)
Statistical Analysis 1: Comparison: TBPM-PI-HBr 600 mg vs Ertapenem 1 g; Test type: Other; p = 0.736, Log Rank

26. Secondary Outcome: Rate of Clinical Relapse at the LFU Days in the Micro-ITT Population
Description: Clinical relapse is participants who met criteria for clinical cure at TOC, but new signs and symptoms of cUTI or AP are present at the LFU Visit and the subject requires antibiotic therapy for the cUT. Clinical cure is defined as complete resolution or significant improvement of signs and symptoms of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted.
Time Frame: Day 25 (LFU)
Population: Micro-ITT population included all randomized participants with a confirmed diagnosis of cUTI or AP and a positive Screening urine culture defined as growth of one or two uropathogens at ≥10^5 CFU/mL and/or positive Screening blood culture with isolation of one or more uropathogens.
Measure: Number; unit: percentage of participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
percentage of participants | 2.7 | 3.6

27. Secondary Outcome: Rates Of Superinfection And New Infection In The Micro-ITT Population
Description: Superinfection was isolation of a new uropathogen at ≥105 CFU/mL (other than the original Baseline pathogen[s] from blood and/or urine) from a urine culture that was accompanied by clinical signs and symptoms of infection requiring alternative antimicrobial therapy (e.g., the participant was assessed by the investigator as a clinical failure) during the period up to and including EOT. New infection was isolation of a new uropathogen at ≥105 CFU/mL (other than the original baseline pathogen[s] from blood and/or urine) from a urine culture that was accompanied by clinical signs and symptoms of infection requiring alternative antimicrobial therapy (e.g., the participant was assessed by the Investigator as a clinical failure) in the period after EOT.
Time Frame: Day 25 (LFU)
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
Number analyzed (Participants) | 449 | 419
percentage of participants
  Superinfection | 0.2 | 2.1
  New Infection | 1.1 | 1.9

28. Secondary Outcome: Apparent Volume of Distribution (Vss) at Steady State in TBPM-PI-HBr Recipients in the Pharmacokinetic (PK) Population
Time Frame: Predose and post-dose at 0.25h, 0.5h, 1h, 2h, and 8h on Days 1 and 3
Population: PK population included participants treated with at least 1 dose of TBPM-PI-HBr with at least 1 analyzable plasma or urine PK sample. The data is reported only for TBPM-PI-HBr arm.
Measure: Mean (Full Range); unit: Liters (L)
Arm/Group | TBPM-PI-HBr 600 mg
Number analyzed (Participants) | 29
Liters (L)
  Day 1 | 75.5 [49.5 to 89.9]
  Day 3 | 75.5 [49.5 to 89.9]

29. Secondary Outcome: Cmax in TBPM-PI-HBr Recipients in the PK Population
Time Frame: Predose and post-dose at 0.25h, 0.5h, 1h, 2h, and 8h on Days 1 and 3
Population: as for outcome 28
Measure: Mean (Full Range); unit: microgram per milliliter (μg/mL)
Arm/Group | TBPM-PI-HBr 600 mg
Number analyzed (Participants) | 29
microgram per milliliter (μg/mL)
  Day 1 | 7.01 [2.05 to 17.2]
  Day 3 | 7.21 [2.11 to 18.8]

30. Secondary Outcome: Area Under Curve (AUC 0-24) in TBPM-PI-HBr Recipients in the PK Population
Time Frame: Predose and post-dose at 0.25h, 0.5h, 1h, 2h, and 8h on Days 1 and 3
Population: as for outcome 28
Measure: Mean (Full Range); unit: microgram.hour per milliliter (μg•h/mL)
Arm/Group | TBPM-PI-HBr 600 mg
Number analyzed (Participants) | 29
microgram.hour per milliliter (μg•h/mL)
  Day 1 | 65.5 [27.6 to 243]
  Day 3 | 74.6 [27.6 to 318]

31. Secondary Outcome: Minimum Concentration (Cmin) in TBPM-PI-HBr Recipients in the PK Population
Time Frame: Predose and post-dose at 0.25h, 0.5h, 1h, 2h, and 8h on Days 1 and 3
Population: PK population included subjects treated with at least 1 dose of TBPM-PI-HBr with at least 1 analyzable plasma or urine PK sample. The data is reported only for TBPM-PI-HBr arm.
Measure: Mean (Full Range); unit: μg/mL
Arm/Group | TBPM-PI-HBr 600 mg
Number analyzed (Participants) | 29
μg/mL
  Day 1 | 0.706 [0.000913 to 4.89]
  Day 3 | 1.17 [0.000877 to 8.44]

32. Secondary Outcome: Systemic Clearance (CL) in TBPM-PI-HBr Recipients in the PK Population
Time Frame: Predose and post-dose at 0.25h, 0.5h, 1h, 2h, and 8h on Days 1 and 3
Population: as for outcome 31
Measure: Mean (Full Range); unit: Litre per hour (L/h)
Arm/Group | TBPM-PI-HBr 600 mg
Number analyzed (Participants) | 29
Litre per hour (L/h)
  Day 1 | 31.6 [5.65 to 65.3]
  Day 3 | 31.6 [5.65 to 65.3]

ADVERSE EVENTS:
Time Frame: From the first dose of administration up to Day 25 post-treatment ± 2 days (up to approximately 27 days)
Description: Safety analysis population included all randomized participants who received any amount of study drug.
Arm/Group | TBPM-PI-HBr 600 mg | Ertapenem 1 g
All-Cause Mortality (participants affected / at risk) | 0/685 | 0/687
Serious Adverse Events (participants affected / at risk) | 14/685 | 12/687
Other Adverse Events (participants affected / at risk) | 39/685 | 30/687
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TBPM-PI-HBr 600 mg (N=685) | Ertapenem 1 g (N=687)
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Cyst (General disorders) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Clostridium test positive (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized tonic-clonic seizure (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TBPM-PI-HBr 600 mg (N=685) | Ertapenem 1 g (N=687)
Diarrhoea (Gastrointestinal disorders) | 39 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 45 days to preserve intellectual property

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT03788967/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT03788967/SAP_001.pdf